CLINICAL TRIAL: NCT06407843
Title: Effects of Schroth Method on Curve Magnitude, Endurance of Lumbar Extensors, and Chest Mobility in Idiopathic Scoliosis
Brief Title: Effects of Schroth Method in Idiopathic Scoliosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/RCR&AHS/23/07105
Record Dates: First submitted 2024-05-06; First posted 2024-05-09 (Actual); Last update posted 2025-03-12 (Actual); Status verified 2025-03

CONDITIONS: Idiopathic Scoliosis
Keywords: Cobb angle; Chest mobility; Idiopathic scoliosis; Lumbar muscle endurance; Schroth Exercise therapy

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Schroth Method (Experimental): In addition to regular physical therapy, this group will engage in Schroth exercises therapy (SET). These regular workouts will include breathing exercises, posture training, spinal flexibility exercises, and stretching activities (especially for the muscles on the concave side of the curve). Patients were positioned asymmetrically to optimize trunk rectification. These exercises will include spinal elongation, de-flexion, stretching, de-rotation, and strengthening. To provide passive support and correct posture during the SET, long poles, foam blocks, and rice sacks were employed. Ten sessions total (30 minutes each, five days a week) will be conducted.
  Interventions: Other: Schroth Method; Other: Regular Physical Therapy
- Regular Physical Therapy (Experimental): This Group will engage in independent routine physical therapy (RPT). Stretching exercises (especially for the muscles on the concave side of the curve) will be part of these regular workouts. The patient will be actively taught standard upper extremity range-of-motion exercises. Without using any creams or lotions, myofascial release (MFR) procedures will be applied straight to the skin. To assist avoid back discomfort, pressure will be administered to the restricted area for 90-120 seconds in order to release the tissue. Twice day, perform 10 repetitions of a 5-second hold while supine pelvic tilt, twice. The same protocol will be followed for the cat and camel, double-leg abdominal presses, and superwoman exercises. There will be breathing exercises including thoracic expansion and diaphragmatic breathing.
  Interventions: Other: Regular Physical Therapy

INTERVENTIONS:
Other: Schroth Method — In addition to regular physical therapy, Group A will engage in Schroth exercises therapy (SET). These regular workouts will include breathing exercises, posture training, spinal flexibility exercises, and stretching activities (especially for the muscles on the concave side of the curve). Ten sessions total (30 minutes each, five days a week) will be conducted.
  Arms: Schroth Method
Other: Regular Physical Therapy — Stretching exercises (especially for the muscles on the concave side of the curve) will be part of these regular workouts. Twice day, perform 10 repetitions of a 5-second hold while supine pelvic tilt, twice. Ten sessions total (30 minutes each, five days a week) will be conducted.

SUMMARY:
A spinal malformation called scoliosis typically manifests in the first two decades of life. It is defined as a lateral curvature of the spine larger than 10, which can be identified by an x-ray using the Cobb angle. Clinically, idiopathic scoliosis is defined as a spinal curvature in the coronal plane of more than 10 degrees. It accounts for 85% of nearly all scoliosis cases. It is advised that patients with curves less than 45° get nonoperative care. The Schroth technique is mostly utilized in the treatment of scoliosis. This technique uses a physiotherapeutic approach to stretch and strengthen any weak muscles. The study's objective is to ascertain how the Scroth method affects the size of the curve, the lumbar extensors' endurance, and the mobility of the chest in cases with idiopathic scoliosis.

The present research will employ a randomized control trial design, with data sourced from the Children Hospital and Institute of Child Health in Lahore, as well as the Pakistan Society for the Rehabilitation of the Disabled, Lahore (PSRD). Thirty-two patients total will be randomly assigned to two equal groups for the study. The study's inclusion criteria will include any patient with idiopathic scoliosis who is between the ages of 9 and 17 and has a Cobb angle between 10˞ and 26˞, regardless of gender. The study will not include any patients with neurological conditions, other orthopedic conditions, surgery histories involving the spine, severe systemic disorders, psychological conditions, or neuromuscular disorders. The experimental group will engage in both routine physical therapy (RPT) and Schroth exercise therapy (SET), while the control group will only receive normal physical treatment. Chest mobility, lumbar extensor endurance, and curve magnitude (Cobb angle) will all be examined. The Sorensen test for lumbar muscle endurance, the X-ray for Cobb angle, and the measuring tape for chest mobility will be the instruments utilized to collect data. The data analysis tool of choice will be SPSS 23.00.

DETAILED DESCRIPTION:
Group A: In addition to regular physical therapy, Group A will engage in Schroth exercises therapy (SET). These regular workouts will include breathing exercises, posture training, spinal flexibility exercises, and stretching activities (especially for the muscles on the concave side of the curve). The intensity of the workout program will progressively rise in line with each participant's improved functional ability. Schroth exercises, which are based on kinesthetic and sensorimotor concepts, will include both passive and active posture autocorrection exercises that are performed frequently. Postural motor control will be enhanced by doing corrective motions repeatedly. Strength and endurance training of the postural muscles is another component of Schroth exercises therapy, which aims to enhance the curve, improve the patient's self-image, and lessen pain. Patients were positioned asymmetrically to optimize trunk rectification. The program will consist of activities designed to increase the curvature, muscle strength, and endurance of postural muscles. These exercises will include spinal elongation, de-flexion, stretching, de-rotation, and strengthening. To provide passive support and correct posture during the SET, long poles, foam blocks, and rice sacks were employed. Depending on how well the patient performs the exercises, the intensity of the Schroth exercises will be gradually raised by modifying the patient's position, varying the number of sets and repetitions of the exercises, and reducing the quantity or degree of passive support. Ten sessions total (30 minutes each, five days a week) will be conducted.

Group B: Group B will engage in independent routine physical therapy (RPT). Stretching exercises (especially for the muscles on the concave side of the curve) will be part of these regular workouts. The patient will be actively taught standard upper extremity range-of-motion exercises. Without using any creams or lotions, myofascial release (MFR) procedures will be applied straight to the skin. To assist avoid back discomfort, pressure will be administered to the restricted area for 90-120 seconds in order to release the tissue. Twice day, perform 10 repetitions of a 5-second hold while supine pelvic tilt, twice. The same protocol will be followed for the cat and camel, double-leg abdominal presses, and superwoman exercises. There will be breathing exercises including thoracic expansion and diaphragmatic breathing.

ELIGIBILITY:
Inclusion Criteria:

* Ages 9 to 17
* Both genders will be included.
* X-rays will show idiopathic scoliosis with Cobb Angle 10-26.

Exclusion Criteria:

* Any type of cerebral illness
* Any other skeletal issue
* Spine procedure history
* Severe systemic illness

Ages: 9 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 32 (Actual)
Dates: Start 2024-05-15 (Actual); Primary Completion 2024-08-05 (Actual); Study Completion 2024-10-15 (Actual)

PRIMARY OUTCOMES:
Cobb angle using X-rays to determine curve magnitude | Baseline and 2 weeks
  By measuring the end vertebra tilt angles, one may determine the Cobb angle, which is the curve magnitude that is the sum of the upper and lower end vertebra tilt angles.
  Just identifying the two end vertebrae and measuring the tilt angles will yield an accurate and quick computation of the Cobb angle. The tilt angle method's measurement steps are as follows:
  1. Sketch the connecting line between the upper and lower vertebral endplates on the film.
  2. Determine the upper and lower endplate tilt angles.
  3. To calculate the Cobb angle, add the two measured findings.

SECONDARY OUTCOMES:
Sorenson test to measure Lumbar extensor muscle | Baseline and 2 weeks
  To evaluate the lumbar extensor muscles' isometric endurance, the Sorensen test will be employed. The duration of the test determines how long the subjects' lumbar muscles can withstand an isometric contraction. The test is discontinued as a precaution after the maximumne position and doing trunk extension.While the second therapist monitors the accuracy of the test and maintains track of time, one therapist holds the participant's lower extremities. Two warnings later, the experiment is discontinued. Following the test, time is calculated to the nearest twenty seconds, with a precision of 0.1 seconds.
Measuring tape to measure chest Mobility | Baseline and 2 weeks
  At rest and during a maximal inhalation and expiration, the chest mobility will be measured using a non-stretch measuring tape at the level of the xyphoide.

CONTACTS AND LOCATIONS:
Overall Officials: Anna Zaheer, MSPT-(NMPT), Study Chair — Riphah International University Lahore; Mowadat Zahra, MSPT-(PPT), Principal Investigator — Riphah International University, Lahore
Locations (1):
- pakistan Society for the Rehabilitaion of Disables, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Strukčinskaitė V, Raistenskis J, Šidlauskienė A, Strukčinskienė B, Griškonis S. EFFECTS OF THE SCHROTH METHOD FOR TRUNK MUSCLES'STATIC ENDURANCE AND SPINE MOBILITY IN GIRLS WITH IDIOPATHIC SCOLIOSIS. Health sciences. 2017;27(5):71-5.
- [Background] Athawale V, Phansopkar P, Darda P, Chitale N, Chinewar A. Impact of Physical Therapy on Pain and Function in a Patient With Scoliosis. Cureus. 2021 May 26;13(5):e15261. doi: 10.7759/cureus.15261. PMID 34188999
- [Background] Blevins K, Battenberg A, Beck A. Management of Scoliosis. Adv Pediatr. 2018 Aug;65(1):249-266. doi: 10.1016/j.yapd.2018.04.013. Epub 2018 Jun 12. No abstract available. PMID 30053928
- [Background] Kocaman H, Bek N, Kaya MH, Buyukturan B, Yetis M, Buyukturan O. The effectiveness of two different exercise approaches in adolescent idiopathic scoliosis: A single-blind, randomized-controlled trial. PLoS One. 2021 Apr 15;16(4):e0249492. doi: 10.1371/journal.pone.0249492. eCollection 2021. PMID 33857180
- [Background] Park J, So WY. The Effect of the Schroth Rehabilitation Exercise Program on Spinal and Feet Alignment in Adolescent Patients with Idiopathic Scoliosis: A Pilot Study. Healthcare (Basel). 2022 Feb 20;10(2):398. doi: 10.3390/healthcare10020398. PMID 35207011